CLINICAL TRIAL: NCT00956462
Title: Topical Steroids Versus Topical Non-steroidal Anti-inflammatory Drugs Following Ahmed Valve Glaucoma Drainage Device Surgery
Brief Title: Steroids Versus Non-steroidal Anti-inflammatory Drugs Following Glaucoma Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: University Health Network, Toronto, University Health Network, toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Trope2009
Record Dates: First submitted 2009-07-17; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-07

CONDITIONS: Glaucoma
Keywords: intraocular pressure; Ahmed valve; NSAIDS; steroids
MeSH Terms: conditions — Glaucoma | interventions — Ketorolac; Anti-Inflammatory Agents, Non-Steroidal; Steroids; Ketorolac Tromethamine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NSAID (Experimental)
  Interventions: Drug: Ketorolac (NSAID) versus Dexamethasone (steroid)
- Steroids (Active Comparator)
  Interventions: Drug: Ketorolac (NSAID) versus Dexamethasone (steroid)

INTERVENTIONS:
Drug: Ketorolac (NSAID) versus Dexamethasone (steroid) — Topical NSAID versus topical steroid after implantation of glaucoma drainage device
  Other Names: Acular (NSAID); Maxidex (steroid)

SUMMARY:
This study aims to evaluate the eye pressure response to non-steroidal anti-inflammatory eye drops as compared to steroid eye drops following glaucoma surgery.

DETAILED DESCRIPTION:
Glaucoma is a chronic disease of the eye which results in gradual loss of nerve fibres, resulting in visual loss. The mainstay of treatment is reduction of intraocular pressure (IOP), which has been shown to preserve vision, and glaucoma surgery aims to achieve this. One type of surgery involves insertion of a glaucoma drainage device (GDD). Following surgery steroid eye drops are commonly used in order to reduce the inflammation that occurs as a result of the surgery. However, a common side effect of steroid eye drops is a rise in eye pressure. Non-steroidal anti-inflammatory drugs (NSAID) eye drops do not have this side effect and are used as an alternative to steroids following other types of eye surgery. Use of NSAID drops following GDD surgery may result in improved eye pressure. This study aims to evaluate the eye pressure response to NSAID eye drops following GDD surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 85 years of age
2. Undergoing glaucoma drainage device surgery

Exclusion criteria

1. Unable to consent
2. Undergoing combined GDD and cataract surgery
3. Patients with conditions requiring additional anti-inflammatory medications e.g., uveitic glaucoma, previous corneal transplant
4. Patients with prior history of corneal ulceration
5. Breast-feeding (nursing) mothers
6. Pregnant or planning to become pregnant during the trial period
7. Allergic to Ketorolac Tromethamine, or had an allergic-type reaction to acetylsalicylic acid or other non-steroidal anti-inflammatory drugs used for pain relief or arthritis

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | Six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Graham Trope, MD FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Graham Trope, Toronto, Ontario, Canada